CLINICAL TRIAL: NCT02498067
Title: rPlan Multimedia Dual Protection Intervention to Reduce Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB14-0379
Record Dates: First submitted 2015-06-16; First posted 2015-07-15 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Sexually Transmitted Infection
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Participants will complete a 10-15 minute questionnaire . After completing the questionnaire, a research assistant (RA) will provide a brief orientation to the rPlan app and use the rPlan app for up to 15 minutes. After viewing rPlan, participants will be asked a series of questions regarding the app's usability, helpfulness, and content appropriateness (10 min). The participant will also be given an STI test.
  Interventions: Behavioral: rPlan dual protection waiting room app intervention

INTERVENTIONS:
Behavioral: rPlan dual protection waiting room app intervention

SUMMARY:
The investigators will develop a digital application (app)-"rPlan dual protection" (rPlan)-to be used in the clinic waiting room prior to a gynecological and/or contraceptive visit. The goal of this research is to develop the app and conduct a feasibility, acceptability and effectiveness assessment of rPlan to examine improvement in dual protection behaviors, enhancement of contraceptive adherence and continuation, increase of condom use and decrease of sexually transmitted infection (STI) and human immunodeficiency virus(HIV) infection. The research will consist of baseline activities and a 12-week in-clinic survey and STI test, as well as a retrospective chart review.

DETAILED DESCRIPTION:
Using the investigators' experience in digital media, behavior theory, client-centered interventions, and family planning, the investigators will develop a digital application ("app")-rPlan-to be used in the clinic waiting room prior to a gynecological and/or contraceptive visit. The goal of this research is to develop the app and conduct a feasibility, acceptability and effectiveness assessment of rPlan.

This study will develop rPlan, a three-part intervention that includes a precounseling app that promotes dual protection, motivational interviewing-informed counseling, and concomitant printed educational materials.

The research will proceed in two phases. In Phase I, the investigators will assemble a 10-member stakeholder advisory team to enhance the PreCounselor app to focus on dual protection, train reproductive health counselors in motivational interviewing, and create concomitant printed educational materials. In Phase II, the feasibility, acceptability, and effectiveness of the intervention will be assessed. The specific aims are to:

Aim 1: Develop the rPlan intervention by (1) enhancing the pretested PreCounselor app to focus on dual protection, (2) training reproductive health counselors, and (3) creating concomitant printed educational materials.

Aim 2: Conduct a pre/post feasibility, acceptability, and effectiveness assessment of rPlan to examine improvement in dual protection behaviors, enhancement of contraceptive adherence and continuation, increase of condom use, and decrease of STI/HIV infection.

The primary outcome is engagement in dual protection (either using a condom with another effective method, or using a condom alone), which will be measured via patient report at 12 weeks post enrollment. The secondary outcomes are contraceptive adherence/uptake (measured at 12 weeks post enrollment), contraceptive decisional balance/self-efficacy (measured at 12 weeks post enrollment), contraceptive effectiveness knowledge, and STI infection (12 weeks post enrollment).

The research will consist of baseline activities as well as a 12-week in-clinic survey and STI test, and a retrospective chart review to capture interceding visits (e.g., initial contraceptive method selection, method switching, etc.) and diagnoses (e.g., pregnancy, STI/HIV).

ELIGIBILITY:
Inclusion Criteria:

* African American (AA) female and sexually active with a male partner(s) within the past 6 months;
* Age 15-24 years;
* Initiating contraception;
* English speaking

Exclusion Criteria:

* Not currently pregnant or intending pregnancy within the next 6 months
* Not currently using the implant or intrauterine device (IUD).

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago, Dept. of OBGYN
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants completed a 10-15 minute questionnaire of sociodemographics, and contraceptive behaviors, self-efficacy, knowledge, and attitudes. Afterwards, a research assistant (RA) provided them with a brief orientation to the rPlan app. Participants then used the rPlan app for up to 15 minutes. After viewing rPlan, participants were asked a series of questions regarding the app's usability, helpfulness, and content appropriateness (10 min). The participant then entered into a 10-minute motivational interviewing session with an RA that addressed ambivalence about using and maintaining a contraceptive method of interest. Afterwards, participants entered into their visit with a provider and completed an STI test.
  3-month followup: Participants returned to the clinic site and completed a questionnaire of contraceptive behaviors, knowledge, and attitudes.
Period: Overall Study
Arm/Group | Intervention
Started | 104
Completed | 71
Not Completed | 33
Not completed — Lost to Follow-up | 22
Not completed — Did not meet inclusion criteria | 11

BASELINE CHARACTERISTICS:
Population: Inclusion criteria: Black, assigned female sex at birth, between 15-25 years in age (inclusive), sexually active with at least one male partner in past six months, initiating contraception, not currently pregnant or intending pregnancy within next six months, English speaking, not currently using a LARC method
Groups:
- Intervention: Participants completed a 10-15 minute questionnaire of sociodemographics, and contraceptive behaviors, self-efficacy, knowledge, and attitudes. Afterwards, a research assistant (RA) provided them with a brief orientation to the rPlan app. Participants then used the rPlan app for up to 15 minutes. After viewing rPlan, participants were asked a series of questions regarding the app's usability, helpfulness, and content appropriateness (10 min). The participant then entered into a 10-minute motivational interviewing session with an RA that addressed ambivalence about using and maintaining a contraceptive method of interest. Afterwards, participants entered into their visit with a provider and completed an STI test.
  6 week followup: Participants completed a 15-25 minute phone survey of their contraceptive behaviors, knowledge, and attitudes.
  3-month followup: Participants returned to the clinic site and completed a questionnaire of contraceptive behaviors, knowledge, and attitudes.
Arm/Group | Intervention
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline
  Participants
    number analyzed (Participants) | 93
    <=18 years | 30
    Between 18 and 65 years | 63
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline
  years
    number analyzed (Participants) | 93
    (all) | 20.0 [15 to 25]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline
  Participants
    number analyzed (Participants) | 93
    Female | 93
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline
  Participants
    Black or African American: number analyzed (Participants) | 93
    Black or African American | 93
Relationship Status [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline. 1 participant did not provide data for this measure.
  Participants
    number analyzed (Participants) | 92
    Single | 35
    Dating/Casual partners | 15
    In relationship | 42
Highest Education Completed [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  Participants
    number analyzed (Participants) | 93
    High school diploma or less | 37
    Some college | 44
    College degree or higher | 12
Age at First Sexual Intercourse [Mean (Full Range); unit: years] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  years
    number analyzed (Participants) | 93
    (all) | 16.1 [12 to 23]
Number of Sexual Partners in Lifetime [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline. 1 participant did not provide data for this measure.
  Participants
    number analyzed (Participants) | 92
    1 partner | 17
    2 partners | 17
    3 partners | 13
    4 partners | 15
    5+ partners | 30
Ever Tested Positive for STI? [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  Participants
    number analyzed (Participants) | 93
    Yes | 31
    No | 62
Pregnancy History [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  Participants
    number analyzed (Participants) | 93
    Never been pregnant | 60
    2 pregnancies | 21
    3+ pregnancies | 12
Age at First Pregnancy [Mean (Full Range); unit: years] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline. 60 participants did not provide data for this measure, as they had never been pregnant.
  years
    number analyzed (Participants) | 33
    (all) | 18.1 [15 to 24]
Number of Births [Count of Participants; unit: Participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  Participants
    number analyzed (Participants) | 93
    0 | 61
    1 | 17
    2+ | 15
Number of Living Children [Mean (Full Range); unit: children] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline. 61 participants did not provide data for this measure.
  children
    number analyzed (Participants) | 32
    (all) | 1.5 [1 to 3]
Contraceptive Method Awareness [Number; unit: participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  participants
    Withdrawal: number analyzed (Participants) | 93
    Withdrawal | 74
    Condom: number analyzed (Participants) | 93
    Condom | 81
    Pill: number analyzed (Participants) | 93
    Pill | 71
    Ring: number analyzed (Participants) | 93
    Ring | 59
    Patch: number analyzed (Participants) | 93
    Patch | 54
    Shot: number analyzed (Participants) | 93
    Shot | 66
    Intrauterine device (IUD): number analyzed (Participants) | 93
    Intrauterine device (IUD) | 45
    Implant: number analyzed (Participants) | 93
    Implant | 49
Past Contraceptive Method Use [Number; unit: participants] — Population: 11 participants were excluded from analysis for failing to meet inclusion criteria, i.e., already using a LARC method at baseline.
  participants
    Never used method: number analyzed (Participants) | 93
    Never used method | 1
    Withdrawal: number analyzed (Participants) | 93
    Withdrawal | 52
    Condom: number analyzed (Participants) | 93
    Condom | 69
    Pill: number analyzed (Participants) | 93
    Pill | 46
    Ring | 3
    Patch: number analyzed (Participants) | 93
    Patch | 9
    Shot: number analyzed (Participants) | 93
    Shot | 37
    IUD: number analyzed (Participants) | 93
    IUD | 5
    Implant: number analyzed (Participants) | 93
    Implant | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Recent Dual Method Use
Description: Reported frequency of use of condoms with another contraceptive method in past 3 months
  5 option close-ended question, ranging from 1 - none of the time, to 5 - every time
Time Frame: Baseline, 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 71
score on a scale
  Baseline, pre-app use | 3.17 [1 to 5]
  3-month follow-up | 3.45 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of whether participants' mean reported scores for frequency of dual method use differ between baseline (pre-rPlan) and 3-month follow-up (post-rPlan); Test type: Other; p = .177, t-test, 2 sided — a priori threshold for statistical significance: p<0.05

2. Primary Outcome: Change in Frequency of Recent Condom Use (by Itself, With no Other Method)
Description: Reported frequency of use of condoms alone (without another method) in past 3 months
  5 option close-ended question, ranging from 1 - none of the time, to 5 - every time
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 71
score on a scale
  Baseline (pre-app use) | 3.15 [1 to 5]
  3-month follow-up | 2.93 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of whether participants' mean reported scores for frequency of condom use alone (without another method) differ between baseline (pre-rPlan) and 3-month follow-up (post-rPlan); Test type: Other; p = .318, t-test, 2 sided — a priori threshold for statistical significance: p<.05

3. Secondary Outcome: Change in Consistency of Recent Contraceptive Use
Description: Self-reported answer (yes or no) to whether participants used contraception every time they had sex in the past three months
Time Frame: Baseline, 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample at baseline and the sample retained at followup. 16 of the 71 retained participants did not have sex during the 3-month time period.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Participants will complete a 10-15 minute questionnaire . After completing the questionnaire, a research assistant (RA) will provide a brief orientation to the rPlan app and use the rPlan app for up to 15 minutes. After viewing rPlan, participants will be asked a series of questions regarding the app's usability, helpfulness, and content appropriateness (10 min). The participant will also be given an STI test.
  rPlan dual protection waiting room app intervention
Arm/Group | Intervention
Number analyzed (Participants) | 55
Participants
  Baseline (pre-app use): Yes | 35
  Baseline (pre-app use): No | 20
  3-month follow-up: Yes | 46
  3-month follow-up: No | 9
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of whether participants reported more consistent contraceptive use (i.e., using contraception every time they had sex) between baseline (pre-rPlan) and 3-month follow-up (post-rPlan); Test type: Other; p = .000, t-test, 2 sided — a priori threshold for statistical significance: p<.05

4. Secondary Outcome: Current Main Method of Contraception
Description: Participants' current main method of contraception, by method type: no method or withdrawal, condom, short-term/combined hormonal (pill, patch, shot, ring), Long acting reversible contraception (LARC: IUD or implant)
Time Frame: Baseline, 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up. 1 participant at 3-month follow-up did not give a response.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 71
Participants
  Baseline (pre-app use): No method or withdrawal | 24
  Baseline (pre-app use): Condom | 13
  Baseline (pre-app use): Hormonal, short-term (pill, patch, shot, ring) | 34
  Baseline (pre-app use): LARC (IUD or implant) | 0
  3-month follow-up: number analyzed (Participants) | 70
  3-month follow-up: No method or withdrawal | 15
  3-month follow-up: Condom | 5
  3-month follow-up: Hormonal, short-term (pill, patch, shot, ring) | 31
  3-month follow-up: LARC (IUD or implant) | 19

5. Secondary Outcome: Change in Future Intentions to Use IUD
Description: Participants' self-reported likelihood of using an IUD in the future, on a close-ended 5-point scale ranging from:
  1 - very unlikely, to 5 - very likely
Time Frame: Baseline (pre-app use), Immediately post-app use
Population: 1 participant did not provider data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 92
score on a scale
  Baseline, pre-app use | 2.38 [1 to 5]
  Baseline, immediately post-app use | 2.70 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported likelihood to use an IUD in the future (on a scale ranging from 1- very unlikely, to 5- very likely) before and directly after using the rPlan app; Test type: Other; p = .030, t-test, 2 sided — a priori threshold for statistical significance: p<.05

6. Secondary Outcome: Change in Future Intentions to Use Implant
Description: Participants' self-reported likelihood of using a contraceptive implant in the future, on a close-ended 5-point scale ranging from:
  1 - very unlikely, to 5 - very likely
Time Frame: Baseline (pre-app use), Immediately post-app use
Population: 2 participants did not provide data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 91
score on a scale
  Baseline (pre-app use) | 2.45 [1 to 5]
  Immediately post-app use | 2.66 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported likelihood to use an implant in the future (on a scale ranging from 1- very unlikely, to 5- very likely) before and directly after using the rPlan app; Test type: Other; p = .140, t-test, 2 sided — a priori threshold for statistical significance: p<.05

7. Secondary Outcome: Change in Future Intentions to Use Condoms
Description: Participants' self-reported likelihood of using condoms in the future, on a close-ended 5-point scale ranging from:
  1 - very unlikely, to 5 - very likely
Time Frame: Baseline (pre-app use), Immediately post-app use
Population: 3 participants did not provide data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 90
score on a scale
  Baseline (pre-app use) | 4.22 [1 to 5]
  Immediately post-app use | 4.11 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported likelihood to use condoms in the future (on a scale ranging from 1- very unlikely, to 5- very likely) before and directly after using the rPlan app; Test type: Other; p = .315, t-test, 2 sided — a priori threshold for statistical significance: p<.05

8. Secondary Outcome: Change in Self-efficacy for Contraceptive Use
Description: Participants' self-reported contraceptive self-efficacy, on a close-ended 5-point scale ranging from 1 - not at all confident, to 5 - extremely confident, between baseline (pre-rPlan) and 3-month follow-up
Time Frame: Baseline, 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up.
  4 retained participants did not provide data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 67
score on a scale
  Baseline (pre-rPlan) | 3.93 [1 to 5]
  3-month follow-up | 3.71 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported contraceptive self-efficacy (on a scale ranging from 1- not at all confident, to 5- extremely confident) before and 3 months after engaging in rPlan; Test type: Other; p = .028, t-test, 2 sided — a priori threshold for statistical significance: p<.05

9. Secondary Outcome: Change in Self-efficacy for Condom Use
Description: Participants' self-reported condom self-efficacy, on a close-ended 5-point scale ranging from 1 - not at all confident, to 5 - extremely confident, between baseline (pre-rPlan) and 3-month follow-up
Time Frame: Baseline (pre-rPlan), 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up.
  3 retained participants did not provide data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 68
score on a scale
  Baseline (pre-rPlan) | 3.64 [1 to 5]
  3-month follow-up | 3.65 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported condom use self-efficacy (on a scale ranging from 1- not at all confident, to 5- extremely confident) before and 3 months after engaging in rPlan; Test type: Other; p = .918, t-test, 2 sided — a priori threshold for statistical significance: p<.05

10. Secondary Outcome: Results of STI Test
Description: Results of sexually transmitted infection (STI) test, at baseline and 3 months
Time Frame: Baseline, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 93
Participants
  Baseline: Positive | 8
  Baseline: Negative | 68
  Baseline: None ordered/Missing | 17
  3-month follow-up: Positive | 0
  3-month follow-up: Negative | 63
  3-month follow-up: None ordered/Missing | 30

11. Secondary Outcome: Change in Number of Recent Sexual Partners
Description: Self-reported number of sexual partners in the past three months (for those who were sexually active)
Time Frame: Baseline, 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up.
  21 retained participants did not provide data for this measure.
Measure: Mean (Full Range); unit: number of sexual partners
Arm/Group | Intervention
Number analyzed (Participants) | 50
number of sexual partners
  Baseline | 1.40 [1 to 4]
  3-month follow-up | 1.24 [1 to 4]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' self-reported number of sexual partners in the past 3 months (for those were sexually active) between baseline and 3-month follow-up; Test type: Other; p = .209, t-test, 2 sided — a priori threshold for statistical significance: p<.05

12. Secondary Outcome: Change in Negative Condom Attitudes
Description: Participants' self-reported degree to which they endorse negative condom attitudes (Brown, 1984), on a close-ended 5-point scale ranging from 1 - strongly disagree, to 5 - strongly agree, between baseline (pre-rPlan) and 3-month follow-up
Time Frame: Baseline, 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up.
  5 retained participants did not provide data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 66
score on a scale
  Baseline (pre-rPlan) | 2.03 [1 to 5]
  3-month follow-up | 1.99 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported degree to which they endorse negative condom attitudes (on a scale ranging from 1- strongly disagree, to 5- strongly agree) before and 3 months after engaging in rPlan; Test type: Other; p = .652, t-test, 2 sided — a priori threshold for statistical significance: p<.05

13. Secondary Outcome: Change in Endorsement of Positive Motivators for Condom Use
Description: Participants' self-reported degree to which they endorse positive motivators for condom use, on a close-ended 5-point scale ranging from 1 - strongly disagree, to 5 - strongly agree, between baseline (pre-rPlan) and 3-month follow-up
Time Frame: Baseline (pre-rPlan), 3 months
Population: Data were analyzed for the 71 of the 93 eligible participants enrolled at baseline who were retained at 3-month follow-up. There were no significant differences in baseline scores between the total eligible sample enrolled at baseline and the sample retained at follow-up.
  1 retained participant did not provide data for this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 70
score on a scale
  Baseline (pre-rPlan) | 4.57 [1 to 5]
  3-month follow-up | 4.63 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' reported degree to which they endorse positive motivators for condom use (on a scale ranging from 1- strongly disagree, to 5- strongly agree) before and 3 months after engaging in rPlan; Test type: Other; p = .498, t-test, 2 sided — a priori threshold for statistical significance: p<.05

14. Secondary Outcome: Change in Negative Contraceptive Attitudes
Description: Participants' self-reported importance of negative contraceptive attitudes (Galavotti et al., 1995) in their decision to use contraception, on a close-ended 5-point scale ranging from 1 - not at all important, to 5 - extremely important, between baseline (pre-rPlan) and 3-month follow-up
Time Frame: Baseline (pre-rPlan), 3 months
Population: as for outcome 8
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 67
score on a scale
  Baseline (pre-rPlan) | 2.20 [1 to 5]
  3-month follow-up | 2.20 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' rated importance of negative contraceptive attitudes on their decision to use contraception (on a scale ranging from 1- not at all important, to 5- extremely important) before and 3 months after engaging in rPlan; Test type: Other; p = .977, t-test, 2 sided — a priori threshold for statistical significance: p<.05

15. Secondary Outcome: Change in Endorsement of Positive Motivators for Contraceptive Use
Description: Participants' self-rated importance of positive motivators for contraceptive use (Galavotti et al., 1995) in their decision to use contraception, on a close-ended 5-point scale ranging from 1 - not at all important, to 5 - extremely important, between baseline (pre-rPlan) and 3-month follow-up
Time Frame: Baseline (pre-rPlan), 3 months
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 70
score on a scale
  Baseline (pre-rPlan) | 4.61 [1 to 5]
  3-month follow-up | 4.64 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of participants' rated importance of positive motivators for contraceptive use on their decision to use contraception (on a scale ranging from 1- not at all important, to 5- extremely important) before and 3 months after engaging in rPlan; Test type: Other; p = .673, t-test, 2 sided — a priori threshold for statistical significance: p<.05

16. Secondary Outcome: Change in Contraceptive Effectiveness Knowledge
Description: Percentage of participants who correctly answered questions of which contraceptive methods were more effective at preventing pregnancy, between baseline (pre-app use) and 3-month follow-up
Time Frame: Baseline (pre-app use), 3 months
Population: as for outcome 13
Measure: Number; unit: percentage who answered correctly
Arm/Group | Intervention
Number analyzed (Participants) | 70
percentage who answered correctly
  Baseline (pre-rPlan): Pills vs condoms, % correct | 31.4
  Baseline (pre-rPlan): IUD vs shot, % correct | 35.7
  3-month follow-up: Pills vs condoms, % correct | 16.9
  3-month follow-up: IUD vs shot, % correct | 25.7
Statistical Analysis 1: Comparison: Intervention; Paired samples t-test comparison of proportion of participants who provided correct answers to whether pills or condoms are more effective at preventing pregnancy, before and 3 months after engaging in rPlan; Test type: Other; p = .049, t-test, 2 sided — a priori threshold for statistical significance: p<.05
Statistical Analysis 2: Comparison: Intervention; Paired samples t-test comparison of proportion of participants who provided correct answers to whether the IUD or shot is more effective at preventing pregnancy, before and 3 months after engaging in rPlan; Test type: Other; p = .265, t-test, 2 sided — a priori threshold for statistical significance: p<.05

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 0/104

LIMITATIONS AND CAVEATS:
Loss of participants to follow-up, missing STI results for 15 participants. No control arm, so cannot infer the independent effects of the rPlan intervention on behavior, self-efficacy, attitude, and knowledge outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT02498067/Prot_SAP_000.pdf